CLINICAL TRIAL: NCT00388544
Title: A Prescription for Enhancing Resident Quality of Life
Brief Title: Enhancing Quality of Life for Nursing Home Residents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Ann Kolanowski, Professor of Nursing, Penn State University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 19150; R01NR008910 (NIH); R01NR008910-01A1 (NIH)
Record Dates: First submitted 2006-10-13; First posted 2006-10-17 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Functional Status

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Behavioral: Activity matched to interest
- 2 (Experimental)
  Interventions: Behavioral: Activity matched to function
- 3 (Experimental)
  Interventions: Behavioral: Activity matched to both interest and function
- 4 (No Intervention): Recreational activities are not tailored to either style of interest or function

INTERVENTIONS:
Behavioral: Activity matched to interest — Recreational activities are tailored to subject's style of interest
  Arms: 1
Behavioral: Activity matched to function — Recreational activities are tailored to subjects physical and cognitive functioning
  Arms: 2
Behavioral: Activity matched to both interest and function — Recreational activities are tailored to both style of interest and physical and cognitive functioning.
  Arms: 3

SUMMARY:
Many persons with dementia exhibit behaviors that caregivers find difficult to manage. The purpose of this study is to test the effectiveness of individualized recreational activities for reducing agitation and passivity in persons with dementia.

DETAILED DESCRIPTION:
Most persons with dementia exhibit behavioral symptoms, such as agitation and passivity, at some time in the course of their illness. These behaviors are a source of caregiver burden and often precipitate nursing home placement. There are a number of drugs that can be used to treat these behaviors, but they are costly and have serious adverse effects in a sizable number of people. Non-drug interventions, such as recreational activities, are recommended as the first line of treatment for behavioral symptoms. However, we don't know which activities are most effective for individual residents. The "one size fits all" approach has not been very effective. We are testing an approach that individualizes activities for residents based on their personality style of interest and functional level. We anticipate that this approach will be more effective for reducing behavioral symptoms than routine activities given to all residents. Consenting residents are assessed for personality and functional level and are videotaped during a baseline period and during activities so we can reliably measure behaviors, affect and engagement.

ELIGIBILITY:
Inclusion Criteria:

* English speaking; diagnosis of dementia; a willing informant who knows the subject well and who can provide past personality and other data; a stable dose of any psychoactive drug from pre-baseline through final observation; and presence of agitation or passivity.

Exclusion Criteria:

* delirium or an unstable medical condition; history of Parkinson's disease, Huntington's disease, seizure disorder, stroke, alcoholism, drug abuse, head trauma with loss of consciousness, or psychiatric illness preceding the onset of memory loss; severe vision or hearing impairment; and receiving a new psychoactive medication within the past 30 days.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 128 (Actual)
Dates: Start 2005-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Agitation | During activity intervention, random times outside of activity intervention (during the intervention period), and one week post intervention period
Passivity | During activity intervention, random times outside of activity intervention (during the intervention period), and one week post intervention period

SECONDARY OUTCOMES:
Mood | During activity intervention, random times outside of activity intervention (during the intervention period), and one week post intervention period
Affect | During activity intervention, random times outside of activity intervention (during the intervention period), and one week post intervention period
Engagement | During activity intervention, random times outside of activity intervention (during the intervention period), and one week post intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Ann Kolanowski, PhD, RN, Principal Investigator — Penn State University
Locations (1):
- Nursing homes in Central and Northeast Pennsylvania, University Park, Pennsylvania, United States

REFERENCES:
- [Background] Fick DM, Kolanowski AM, Waller JL, Inouye SK. Delirium superimposed on dementia in a community-dwelling managed care population: a 3-year retrospective study of occurrence, costs, and utilization. J Gerontol A Biol Sci Med Sci. 2005 Jun;60(6):748-53. doi: 10.1093/gerona/60.6.748. PMID 15983178
- [Background] Kolanowski AM, Litaker M, Buettner L. Efficacy of theory-based activities for behavioral symptoms of dementia. Nurs Res. 2005 Jul-Aug;54(4):219-28. doi: 10.1097/00006199-200507000-00003. PMID 16027564
- [Background] Kolanowski A, Litaker M. Social interaction, premorbid personality, and agitation in nursing home residents with dementia. Arch Psychiatr Nurs. 2006 Feb;20(1):12-20. doi: 10.1016/j.apnu.2005.08.006. PMID 16442470
- [Background] Kolanowski A, Buettner L, Litaker M, Yu F. Factors that relate to activity engagement in nursing home residents. Am J Alzheimers Dis Other Demen. 2006 Jan-Feb;21(1):15-22. doi: 10.1177/153331750602100109. PMID 16526585
- [Background] Kolanowski A, Fick D, Waller JL, Ahern F. Outcomes of antipsychotic drug use in community-dwelling elders with dementia. Arch Psychiatr Nurs. 2006 Oct;20(5):217-25. doi: 10.1016/j.apnu.2006.04.004. PMID 17010825
- [Background] Yu F, Kolanowski AM, Litaker M. The association of physical function with agitation and passivity in nursing home residents with dementia. J Gerontol Nurs. 2006 Dec;32(12):30-6. doi: 10.3928/00989134-20061201-05. PMID 17190404
- [Background] Woods CA. Working better with GPs: lessons to be learned from a study of health care networks in the management of diabetes. Clin Exp Optom. 2006 Jan;89(1):1-2. doi: 10.1111/j.1444-0938.2006.00006.x. No abstract available. PMID 16430433
- [Background] Kolanowski A, Buettner L, Moeller J. Treatment fidelity plan for an activity intervention designed for persons with dementia. Am J Alzheimers Dis Other Demen. 2006 Oct-Nov;21(5):326-32. doi: 10.1177/1533317506291074. PMID 17062551
- [Background] Penrod J, Yu F, Kolanowski A, Fick DM, Loeb SJ, Hupcey JE. Reframing person-centered nursing care for persons with dementia. Res Theory Nurs Pract. 2007;21(1):57-72. doi: 10.1891/rtnpij-v21i1a007. PMID 17378465
- [Background] Kolanowski A, Hoffman L, Hofer SM. Concordance of self-report and informant assessment of emotional well-being in nursing home residents with dementia. J Gerontol B Psychol Sci Soc Sci. 2007 Jan;62(1):P20-7. doi: 10.1093/geronb/62.1.p20. PMID 17284553
- [Background] Buettner, L., Kolanowski, A. & Yu, F. (2007). Recreational games: Simple and effective cognitive stimulation programs for residents with dementia in long-term settings. American Journal of Recreation Therapy, 6 (1), 25-30.
- [Background] Kolanowski A, Buettner L. Prescribing activities that engage passive residents. An innovative method. J Gerontol Nurs. 2008 Jan;34(1):13-8. doi: 10.3928/00989134-20080101-08. PMID 18274300
- [Background] Whall AL, Colling KB, Kolanowski A, Kim H, Son Hong GR, DeCicco B, Ronis DL, Richards KC, Algase D, Beck C. Factors associated with aggressive behavior among nursing home residents with dementia. Gerontologist. 2008 Dec;48(6):721-31. doi: 10.1093/geront/48.6.721. PMID 19139246
- [Background] Dettmore D, Kolanowski A, Boustani M. Aggression in persons with dementia: use of nursing theory to guide clinical practice. Geriatr Nurs. 2009 Jan-Feb;30(1):8-17. doi: 10.1016/j.gerinurse.2008.03.001. PMID 19215808
- [Background] Smith, M., Kolanowski, A., Buettner, S., & Buckwalter, K. (accepted). Beyond bingo and painted nails: Meaningful activities for persons with dementia in the nursing home. Annals of Long Term Care.
- [Background] Kolanowski A, Fick DM, Campbell J, Litaker M, Boustani M. A preliminary study of anticholinergic burden and relationship to a quality of life indicator, engagement in activities, in nursing home residents with dementia. J Am Med Dir Assoc. 2009 May;10(4):252-7. doi: 10.1016/j.jamda.2008.11.005. Epub 2009 Jan 9. PMID 19426941
- [Background] Haidet KK, Tate J, Divirgilio-Thomas D, Kolanowski A, Happ MB. Methods to improve reliability of video-recorded behavioral data. Res Nurs Health. 2009 Aug;32(4):465-74. doi: 10.1002/nur.20334. PMID 19434651
- [Background] Lingler JH, Jablonski RA, Bourbonniere M, Kolanowski A. Informed consent to research in long-term care settings. Res Gerontol Nurs. 2009 Jul;2(3):153-61. doi: 10.3928/19404921-20090428-03. Epub 2009 May 29. PMID 20078005
- [Result] Kolanowski A, Litaker M, Buettner L, Moeller J, Costa PT Jr. A randomized clinical trial of theory-based activities for the behavioral symptoms of dementia in nursing home residents. J Am Geriatr Soc. 2011 Jun;59(6):1032-41. doi: 10.1111/j.1532-5415.2011.03449.x. Epub 2011 Jun 7. PMID 21649633